CLINICAL TRIAL: NCT06324630
Title: Implementation of Innovative Food Prescription Programs in Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University at Buffalo (Other)
Collaborators: American Heart Association (Other)
Responsible Party: Principal Investigator, Lucia A Leone, Principal Investigator, University at Buffalo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 24FIM1266996
Record Dates: First submitted 2024-03-04; First posted 2024-03-22 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2024-10

CONDITIONS: Food Preferences; Food Habits
MeSH Terms: conditions — Food Preferences; Feeding Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Produce Prescription Mobile Market (Active Comparator): Usual care control is a produce prescription model prescribed by a clinician, providing funds to purchase 21 servings of fruit and vegetables per person at designated mobile market provider(s).
  Interventions: Other: Produce Prescription Mobile Market
- Produce Prescription Delivery (Experimental): Intervention arm 1 is a healthy food delivery model, wherein the participant receives a customizable produce box providing 21 servings of fruits and vegetables per person.
  Interventions: Other: Produce Prescription Delivery
- Healthy Meal Kit Delivery (Experimental): Intervention arm 2 is a healthy meal kit delivery model providing all ingredients to make 3+ meals with 21 servings of fruits and vegetables, with 6-9 meal options to choose from each week.
  Interventions: Other: Healthy Meal Kit Delivery

INTERVENTIONS:
Other: Produce Prescription Delivery — Fruit and vegetable box delivery
  Arms: Produce Prescription Delivery
Other: Healthy Meal Kit Delivery — Ingredients to cook healthy meals delivered to home
  Arms: Healthy Meal Kit Delivery
Other: Produce Prescription Mobile Market — Voucher to purchase fruits and vegetables at a mobile market
  Arms: Produce Prescription Mobile Market

SUMMARY:
In the USA, about 10% of grown-ups have a hard time finding healthy food, like fruits and vegetables. It's even harder for older grown-ups who might be sick and find it tricky to move around, which makes it tough to get healthy food. The investigators are trying to fix this by testing two new ways to help older people (aged 65 and up) get nutritious food. The investigators are getting lots of help and ideas from older adults to make these ways work the best they can.

The study is happening at the Erie County Medical Center (ECMC) in the East Side of Buffalo, NY, where many African Americans live. This place hasn't been treated fairly, so there aren't many places to buy fresh fruits and vegetables in the local stores. On the ECMC campus, there are three clinics that can help people who can't easily get healthy food. Every participant in our study will be put into one of three programs, each lasting 12 weeks, and they will get food every week.

In the "usual care" program, a doctor writes an order, and the participant gets a voucher to buy more fruits and vegetables at a market or store.

In the "delivery of a produce prescription box" program, a box of fruits and vegetables is brought to the participant's home. The participant can pick what they like online or by calling a helper. If they don't pick, they get a regular box.

In the "delivery of a meal kit box" program, the participant gets the ingredients for three meals in a box. The participant can pick three meals they like online or by calling. If the participant doesn't pick, three meals will be chosen for the participant.

For the second and third programs, participants will get messages to remind the participant when to choose their food, when the time to choose is almost up, and when their food is on its way. If a participant can't use messages or the internet, they can call a helper for support. The investigators believe the study will show that these ways can help older adults who have a hard time getting food to eat more fruits and vegetables. The investigators will also find out which way works best compared to the usual way in the Buffalo, NY area.

DETAILED DESCRIPTION:
Food insecurity in older adults is a complex issue that is growing in scale. This project will compare two innovative produce prescription delivery models against a usual care produce prescription model. The patient population is older adults (aged 65 and over) who have screened positive for food insecurity from one of three primary care clinics in Erie County Medical Center (ECMC). ECMC is located in a medically underserved area of Buffalo, New York, where the majority of the population identifies as African American. Each participant will be randomized to one of the three study arms. Each intervention will give a participant free food (21 servings of fruits and vegetables) weekly for 12 weeks. The usual care arm is receiving access to a mobile market-based produce prescription which can be redeemed at over 10 locations in the city. The first intervention arm will have a fully customizable box of fresh fruits and vegetables delivered to their home. The second intervention arm will be a meal kit delivery box where a participant can choose from 6-9 options weekly. Outcomes compared across arms include enrollment, redemption, and food usage. The investigators will also explore impact of the intervention on fruit and vegetable consumption and related psychosocial behaviors. The investigators will collaborate with an older adult patient advisory group in the development of the two novel interventions and utilize rapid weekly survey feedback to optimize the programs before the end of the 12-week time period. This research will help understand how to best address low utilization rates of food prescription programs with the goal of reducing food insecurity and chronic disease among older adults.

ELIGIBILITY:
Inclusion Criteria:

* Age 65 or over
* English-speaking

Exclusion Criteria:

* Under the age of 65
* Does not speak English
* Cognitively impaired (screen for cognitive function)

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 67 (Actual)
Dates: Start 2024-09-09 (Actual); Primary Completion 2025-02-17 (Actual); Study Completion 2025-02-17 (Actual)

PRIMARY OUTCOMES:
Program Redemption | Measured weekly for duration of 12-week intervention
  Redemption will be measured as the weekly usage of the interventions. Participants will receive an automatic notification after each delivery (or weekly for the usual care arm) and will be asked to confirm that they received their delivery/redeemed their prescription. If they do not initially confirm, they will receive two reminder notifications. Redemption will be measured as the percentage of all 12 deliveries/mobile market visits that are either confirmed via post on the usage survey. Self-report redemption data will also be compared to point-of-sale and delivery software records.

SECONDARY OUTCOMES:
Program Usage | Measured weekly for duration of 12-week intervention
  Usage will be measured in the self-reported weekly text surveys that will ask participants approximately what percentage of the fruits and vegetables that they receive was used by someone in their household: all (coded as 100%), most (coded as 75%), about half (coded as 50%), some (coded as 25%) and none (coded as 0%). Answers from all completed surveys over 12 weeks will be averaged to get a percent usage for each participant.
Program Interest by Consenting to Being Contacted/Voiced Interest to Recruiter | Collected once per eligible individual during approximately 4-week recruitment period
  Program interest will be defined as eligible participants that were referred to the program and expressed interest in the program by providing their information to be contacted about the program. We will collect the number of eligible individuals who agreed to be contacted by researchers after having the program described to them in the clinical setting. We will also collect the number of eligible individuals who were interested in learning more about the project when contacted by the research team for recruitment.
Program Enrollment | Collected once per eligible individual during approximately 4-week recruitment period
  Program enrollment will be measured as the percentage of patients eligible and referred that decide to enroll. Patients who choose not to enroll will be asked to provide more information on why they do not want to enroll.

OTHER OUTCOMES:
Fruit and Vegetable Consumption | Collected at baseline and after 12-week intervention period
  2021 Behavioral Risk Factor Surveillance System Fruit and Vegetable module
Nutrition Security | Collected at baseline and after 12-week intervention period
  Nutrition Security will be measured using a combination of the United States Department of Agriculture Food Security Survey Module, which assesses accessibility and affordability, with the new suite of nutrition security measures that complement the USDA instrument to help capture the remaining pillars of nutrition security (availability, utilization, and stability)
Self-Efficacy to Purchase, Prepare, and Eat Fresh Fruits and Vegetables | Collected at baseline and after 12-week intervention period
  10-point Likert scale (strongly disagree to strongly agree, where a positive score indicates a positive belief) using a selection of items adapted from a study of shoppers where self-efficacy was shown to be correlated with nutrition behaviors.
Barriers to Eating Fruits and Vegetables | Collected at baseline and after 12-week intervention period
  4-point Likert scale (strongly disagree to strongly agree, where a positive score indicates a positive belief) previously tested in lower-income adults which reflects common benefits/barriers found in the literature.
Health Status and Disease Risk | Collected at baseline and after 12-week intervention period
  Health status and disease risk will be measured using the following subscales of the RAND 36-Item Short Form Health Survey (SF-36): 1.) General health: 1 item with a 5-point Likert scale where 1 is excellent and 5 is poor, 4 items using a 5-point Likert scale where 1 is definitely true and 5 is definitely false; 2. Emotional well-being: 5 items with a 6-point Likert scale where 1 is all of the time and 6 is none of the time; and 3.) Social functioning: 1 item with a 5-point Likert scale where 1 is not at all and 5 is extremely and 1 item with a 5-point Likert scale where 1 is all of the time and 5 is none of the time.
Quality of Life in Older Age | Collected at baseline and after 12-week intervention period
  The short version 2 of the validated World Health Organization Quality of Life in Elderly People Scale (WHOQOL-OLD).

CONTACTS AND LOCATIONS:
Overall Officials: Lucia Leone, PhD, Principal Investigator — University at Buffalo; Jill Tirabassi, MPH, MD, Principal Investigator — University at Buffalo
Locations (1):
- University at Buffalo, Buffalo, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data (including data dictionaries) generated within this study (trial) will be provided to the American Heart Association in a de-identified form, to be deposited within the Health Care x Food data repository on the Precision Medicine Platform, and subject to the Precision Medicine Platform Terms and Conditions. Participant data on the Precision Medicine Platform will be collated with data from other studies that are funded by the American Heart Association Health Care x Food initiative, and used by future investigators for analysis.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be made available in alignment with agreed-upon Open Science Policies at the American Heart Association, whereby any factual data that is needed for independent verification of research results must be made freely and publicly available in an AHA-approved repository as soon as possible, and no later than the time of an associated publication or the end of the award period (and any no-cost extension), whichever come first. Data will be available indefinitely.
Access Criteria: Researchers who would like to access the data for the Health Care x Food initiative will be required to create an account on the AHA Precision Medicine Platform and receive approval for their proposed research using the dataset.
  In addition, de-identified participant data will be made available to anyone who wishes to access the data by sending a request to the study PIs via email (lucialeo@buffalo.edu, jilltira@buffalo.edu).